CLINICAL TRIAL: NCT02616380
Title: Real-World Outcome of Adalimumab on Rheumatoid Arthritis Patients in Taiwan
Acronym: ROCKI
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-778
Record Dates: First submitted 2015-11-25; First posted 2015-11-26 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Quality of life (QOL); Work productivity; Rheumatoid arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adalimumab: Participants diagnosed with rheumatoid arthritis who were prescribed adalimumab according to their physician's discretion and routine clinical practice.

SUMMARY:
The study is designed as a prospective, observational study to assess the effect of adalimumab on health-related quality of life (QoL) and work productivity in patients with rheumatoid arthritis (RA) in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of RA as defined by the 1987 revised American College of Rheumatology (ACR) classification criteria and/or the ACR/the European League against Rheumatism (EULAR) 2010 classification criteria (any duration since diagnosis).
* Male or female subjects >= 18 years of age (local definition according to adalimumab label) who is in compliance with eligibility for adalimumab based on the local label.
* Patients with moderate to severe RA defined as Disease Activity Score in 28 Joints (DAS28) Erythrocyte Sedimentation Rate (ESR) or DAS28 C- Reactive Protein (CRP) >3.2
* Biologically treatment naïve and initiated adalimumab at baseline visit
* Availability of clinical data of the previous 12 weeks prior to baseline
* Ability to self-complete patient questionnaires
* Subject must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

Exclusion Criteria:

* Patients who are pregnant or breast feeding at enrolment or wish to become pregnant in the next 24 weeks.
* Participation in any RA-related clinical trial at the time of enrolment, at baseline or at any point during the past 24 weeks prior to baseline
* Patients, who in the clinician's view, may not be able to accurately report their QoL or prior resource utilization
* Patients, who in the clinician's view, may not be able to adhere to adalimumab therapy over 24 weeks.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects receiving Adalimumab with Rheumatoid Arthritis (RA) in Taiwan
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hsieh SC, Tsai PH, Kuo CF, Cheng TT, Lai NS, Lin JC, Lin LH, Tsai CY. Health-related quality of life improvement by adalimumab therapy in patients with rheumatoid arthritis in Taiwan: A nationwide prospective study. J Chin Med Assoc. 2023 Apr 1;86(4):366-374. doi: 10.1097/JCMA.0000000000000889. Epub 2023 Jan 24. PMID 36692418
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred participants with rheumatoid arthritis (RA) were enrolled at 7 sites in Taiwan.
Period: Overall Study
Arm/Group | Adalimumab
Started | 100
Completed | 97
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Heath Assessment Questionnaire - Disability Index [Mean (Standard Deviation); unit: units on a scale] — The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories including dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Patients were asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), where higher scores represent a high-dependency disability.
  units on a scale | 1.06 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 24
Description: The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories representing a comprehensive set of functional activities, including dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Patients were asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), with a higher score representing a high-dependency disability.
Time Frame: Baseline and Week 24
Population: Participants who were still receiving adalimumab at week 24 and with available HAQ-DI data at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 94
units on a scale | -0.44 (0.59)
Statistical Analysis 1: Comparison: Adalimumab; Test type: Other; p < 0.0001, Paired t-test; The mean change was tested with a paired t-test without adjusting for baseline disease severity

2. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Summary and Mental Component Summary Scores at Weeks 12 and 24
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The summary physical health score included the following subscales: physical functioning, role-physical, bodily pain, and general health. The summary mental health score included the following subscales: vitality, social functioning, role-emotional, and mental health.
  Each score ranges from 0 to 100 where higher scores indicate a better quality of life. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline, week 12, and week 24
Population: Participants still receiving adalimumab and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 97
units on a scale
  Physical Component Score at Week 12: number analyzed (Participants) | 95
  Physical Component Score at Week 12 | 5.72 (5.78)
  Physical Component Score at Week 24: number analyzed (Participants) | 93
  Physical Component Score at Week 24 | 8.09 (7.13)
  Mental Component Score at Week 12: number analyzed (Participants) | 95
  Mental Component Score at Week 12 | 3.67 (7.94)
  Mental Component Score at Week 24: number analyzed (Participants) | 93
  Mental Component Score at Week 24 | 5.85 (7.99)
Statistical Analysis 1: Comparison: Adalimumab; Change From Baseline in Physical Component Score at Week 12; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Adalimumab; Change From Baseline in Physical Component Score at Week 24; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: Adalimumab; Change From Baseline in Mental Component Score at Week 12; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: Adalimumab; Change From Baseline in Mental Component Score at Week 24; Test type: Other; p < 0.0001, Paired t-test

3. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension 3-Level (EQ-5D-3L) Index at Weeks 12 and 24
Description: The EQ-5D-5L descriptive system comprises 5 dimensions of health-related quality of life states (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which can take one of three responses. The responses record three levels of severity ('no problems', 'some problems', and 'extreme problems') within a particular EQ-5D-3L dimension. The EQ-5D-3L results were converted into a weighted health state index with scores ranging from approximately 0 (death) to 1 (full health). A positive change from baseline indicates improvement.
Time Frame: Baseline, week 12, and week 24
Population: Participants still receiving adalimumab and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 97
units on a scale
  12 weeks: number analyzed (Participants) | 96
  12 weeks | 0.23 (0.30)
  24 weeks: number analyzed (Participants) | 94
  24 weeks | 0.33 (0.38)
Statistical Analysis 1: Comparison: Adalimumab; Change from Baseline in EQ-5D-3L at 12 weeks; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Adalimumab; Change from Baseline in EQ-5D-3L at 24 weeks; Test type: Other; p < 0.0001, Paired t-test

4. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) at Weeks 12 and 24
Description: The Work Productivity and Activity Impairment (WPAI) questionnaire for general health is a validated tool in RA consisting of 6 questions, based on patient recall of the previous 7 days. WPAI assesses work time missed due to illness (absenteeism), impairment at work due to health (presenteeism), overall work impairment due to health (an aggregate measure of both absenteeism and presenteeism), and total non-occupational activity impairment due to health. WPAI scores are expressed as impairment percentages, with higher scores indicating worse outcomes. A negative change from baseline indicates improvement.
Time Frame: Baseline, week 12, and week 24
Population: Participants still receiving adalimumab and with available data at each time point. Overall work impairment was only assessed in participants who were employed.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Adalimumab
Number analyzed (Participants) | 97
percent impairment
  Overall Work Impairment at Week 12: number analyzed (Participants) | 40
  Overall Work Impairment at Week 12 | -18 (23)
  Overall Work Impairment at Week 24: number analyzed (Participants) | 39
  Overall Work Impairment at Week 24 | -19 (23)
  Activity Impairment at Week 12: number analyzed (Participants) | 95
  Activity Impairment at Week 12 | -14 (22)
  Activity Impairment at Week 24: number analyzed (Participants) | 92
  Activity Impairment at Week 24 | -24 (25)
Statistical Analysis 1: Comparison: Adalimumab; Change From Baseline in Overall Work Impairment at Week 12; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Adalimumab; Change From Baseline in Overall Work Impairment at Week 24; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: Adalimumab; Change From Baseline in Activity Impairment at Week 12; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: Adalimumab; Change From Baseline in Activity Impairment at Week 24; Test type: Other; p < 0.0001, Paired t-test

5. Secondary Outcome: Change From Baseline in HAQ DI Score at Week 12
Description: as for outcome 1
Time Frame: Week 0 and Week 12
Population: Participants who were still receiving adalimumab at week 24 and with available HAQ-DI data at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 96
units on a scale | -0.34 (0.46)
Statistical Analysis 1: Comparison: Adalimumab; Test type: Other; p < 0.0001, Paired t-test; The mean change was tested with a paired t-test without adjusting for baseline disease severity

6. Secondary Outcome: Percentage of Participants Achieving a Clinically Meaningful Improvement on the HAQ-DI at Weeks 12 and 24
Description: The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories representing a comprehensive set of functional activities, including dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Patients were asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), with a higher score representing a high-dependency disability.
  A clinically meaningful improvement was defined as an improvement of -0.22 points or greater in the HAQ-DI score.
Time Frame: Baseline, week 12 and week 24
Population: Participants still receiving adalimumab and with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 97
percentage of participants
  Week 12: number analyzed (Participants) | 96
  Week 12 | 60.4
  Week 24: number analyzed (Participants) | 94
  Week 24 | 59.6

7. Secondary Outcome: Healthcare Resource Utilization: Number of Participants With Visits to Healthcare Professionals for Treatment of Rheumatoid Arthritis
Description: The healthcare resource utilization (HCRU) questionnaire collected data on the healthcare resources used over the course of the study.
Time Frame: 24 weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 100
Participants
  Any healthcare professional | 99
  Rheumatologist | 97
  Traditional medicine | 7
  Orthopaedist | 5
  Rehabilitation medicine | 5
  Family medicine | 3
  Internist | 2
  Emergency department | 1
  Other | 11

8. Secondary Outcome: Healthcare Resource Utilization: Number of Participants Who Underwent Procedures Related to Treatment of Rheumatoid Arthritis
Description: as for outcome 7
Time Frame: 24 weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 100
Participants
  Any Procedure | 95
  Blood Sample Taken | 87
  Chest X-Ray | 27
  Urine Test | 11
  Liverfunction Test | 11
  Electroardiogram | 9
  Hand X-Ray | 5
  Spine X-Ray | 4
  Bone Scan | 3
  Shoulder X-Ray | 1
  Knee X-Ray | 1
  Magnetic Resonance Imaging (MRI) | 1
  Endoscopy | 1
  Tuberculin Skin Test | 1
  Sputum Tests | 1
  Other | 8

9. Secondary Outcome: Healthcare Resource Utilization: Number of Participants With Hospitalization Related to Rheumatoid Arthritis
Description: as for outcome 7
Time Frame: 24 weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 100
Participants | 1

10. Secondary Outcome: Healthcare Resource Utilization: Number of Participants Who Received Concomitant Medications for Rheumatoid Arthritis
Description: as for outcome 7
Time Frame: 24 weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 100
Participants
  Any Concomitant Medication | 100
  Disease Modifying Antirheumatic Drug (DMARD) | 96
  Non-steroidal Anti-inflammatory Drug (NSAID) | 73
  Others | 59

ADVERSE EVENTS:
Time Frame: Up to 34 weeks
Description: The protocol required that all serious adverse events (SAEs) to be actively solicited. Non-serious adverse events were collected as spontaneous reports when the Sponsor was notified.
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 1/100
Other Adverse Events (participants affected / at risk) | 1/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=100)
Hip fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=100)
Allergic reaction (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT02616380/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02616380/SAP_001.pdf